CLINICAL TRIAL: NCT03565497
Title: Engaging Working Memory and Distress Tolerance to Aid Smoking Cessation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic caused human subjects research to shut down and study was unable to restart.
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Michael Otto, Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA046963
Record Dates: First submitted 2018-05-29; First posted 2018-06-21 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wellness Education Control Condition (Placebo Comparator): The wellness education control condition (CC) is modeled after that used in our studies of exercise for smoking cessation, but delivered in an individual format. Content focuses on discussions of a variety of healthy lifestyle topics, such as healthy eating, time management, recommended health screenings, and cancer and cardiovascular prevention. Content is delivered using a combination of lectures, videos, handouts, and discussions while allowing participants to set their own realistic wellness goals, which they can gradually incorporate into their lives.
  Interventions: Behavioral: Wellness Education Control Condition
- Mindfulness Training (MT) (Experimental): Mindfulness training will be adapted for 6 individual sessions;elements include: (1) a body scan designed to teach participants to pay attention to specific parts of their bodies as a strategy to increase attentional capacities/reduce habitual mind-wandering; (2) non-judgmental awareness, and (3) 'awareness of breath' meditation, with an additional focus on helping participants become more aware of the present moment and refrain from habitually engaging in self-related pre-occupations concerning the future or the past.
  Interventions: Behavioral: Mindfulness Training
- Mindfulness Training Plus IE (MT+IE) (Experimental): This condition will mirror the MT condition for the first 4 individual sessions, then for the final 2 individual sessions, MT will be rehearsed under conditions of sensations of anxiety/tension induced by interoceptive exposure procedures (IE).
  Interventions: Behavioral: Mindfulness Training Plus IE

INTERVENTIONS:
Behavioral: Wellness Education Control Condition — As per arm of the same name
  Arms: Wellness Education Control Condition
Behavioral: Mindfulness Training — As per arm of the same name
  Arms: Mindfulness Training (MT)
Behavioral: Mindfulness Training Plus IE — As per arm of the same name
  Arms: Mindfulness Training Plus IE (MT+IE)

SUMMARY:
Specific Aims for this Project Are:

1. To evaluate the ability of two forms of mindfulness training, relative to a control intervention, to engage specific "triple-vulnerability" mechanistic targets that characterize low SES smokers.

   1. The investigators hypothesize that both versions of the mindfulness training will show greater target engagement than the control treatment for mechanistic targets assessed under standard smoking conditions.
   2. The investigators hypothesize that the enhanced mindfulness training, Mindfulness+IE, will show greater target engagement than the other two conditions for mechanistic targets assessed during the nicotine deprivation window.
2. To show that the hypothesized differential target engagement results in differential smoking self-control as evaluated by greater time to lapse, fewer cigarettes smoked, and different smoking topography in the McKee Lapse protocol.
3. To expand and refine the list of SOBC targets by showing the specific relationship between currently identified assays and empirically-validated alternative targets, with attention to showing which of the targeted mechanisms in which contexts are most linked to clinically-relevant outcomes assessed in the McKee protocol, and which offer redundant or non-significant prediction.

DETAILED DESCRIPTION:
This study is designed to evaluate the success of mechanistic target engagement in two specific contexts: under standard smoking conditions and under nicotine deprivation (stress) conditions. After screening, consent, and baseline assessment, participants selected on the basis of inclusion/exclusion criteria will be randomized to one of three intervention conditions: (1) a health-education control condition (CC), (2) a mindfulness training condition (MT), or (3) a mindfulness training condition combined with training applying mindfulness skills in the context of interoceptive exposure (Mindfulness+IE). Following 6 sessions of these interventions, delivered over 3 weeks, participants will then undergo the standard smoking assessment of mechanistic targets. Two days later (and matching the progression to quit-attempt challenges following treatment), participants will undergo the deprivation window assessment (14 hours of smoking abstinence) of these same mechanistic targets, followed by evaluation of lapse behavior and smoking topography in the McKee paradigm to yield: (1) latency to initiate smoking during a monetarily reinforced delay period, (2) the number of cigarettes smoked during a subsequent 60-minute self-administration period, and (3) exploratory analysis of smoking topography: puff volume, puff duration, and inter-puff interval. Participants will be recruited to Boston University through study advertisements targeted to low SES neighborhoods, with attention to health service centers and religious institutions serving low SES individuals.

Following telephone screening for basic eligibility, participants will be scheduled for an informed consent interview and subsequent baseline assessment session. Interventions are to be completed over the subsequent 3 weeks, and post-treatment assessments of the mechanistic targets are scheduled for one-week (standard smoking assessment) and one week + 2 days (deprivation-window assessment) from the last intervention session. For the standard smoking window assessments, participants are asked to smoke .5 hour before the scheduled assessment session. The deprivation-window assessment is scheduled two days later, (for example, scheduled for 12:00 noon, with smoking to cease at 10PM the night before). Upon arrival to the lab, nicotine abstinence will be verified by expired CO levels, as determined by a cut-off of half of the participant's screening session CO concentration or <10 PPM (those failing will be rescheduled). After verification of abstinence, participants will complete assessment of the triple-risk mechanistic target variables. These assessments will be followed by the McKee Lapse protocol: participants will be instructed that over the next 50 min, they will have the option to initiate a cigarette self-administration (smoking) session at any point or to delay initiation in exchange for monetary reinforcement. If participants choose to delay, they will be awarded funds for each 5-minute increment they are able to resist smoking. Once participants choose to end the delay period in order to smoke (or resist smoking for the entire 50 minute delay period), they will then participate in a 60-minute cigarette self-administration session, in which they will be given the choice to either smoke their preferred brand of cigarettes or receive monetary reinforcement for cigarettes not smoked. Participants will be given funds at the beginning of the self-administration session and will lose a portion of the funds for each cigarette smoked. When participants smoke in this protocol, we will use the Clinical Research Support System (CReSS) to measure smoking topography. The reliability and acceptability of use of the portable CReSS device is well documented,88,94 and is recommended over direct observation. Topography data will include puff CO volume, puff duration, and inter-puff interval. Puff level data will be averaged to compute mean topography variables for each participant.

ELIGIBILITY:
Inclusion Criteria:

* be between 18 and 65 years of agehave reported household income of less than 1.5Xpoverty guidelines
* be a regular smoker for at least one year
* report daily smoking (minimum of 5 cigarettes per day and biochemically confirmed via Carbon Monoxide [CO] analysis; > .10ppm CO)
* not be presently engaged in a quit attempt

Exclusion Criteria:

History of psychosis as determined by a brief psychotic screen, pregnancy, nursing mothers, medical conditions that would contraindicate smoking (e.g., current diagnoses of chronic medical diseases including heart disease, chronic obstructive pulmonary disease, or seizure disorders - assessed during telephone prescreen and initial assessment via medical checklist), nicotine use other than cigarette smoking, current use of any pharmacotherapy for smoking cessation, or insufficient command of the English language (i.e., cannot carry on a conversation with an interviewer in the English language or read associated text).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Within one year of completion (publication) of the primary Aims for this project, we will provide de-identified data from this project to interested researchers. The data is to be provided in a SAS file or Excel, with separate documentation of labels/characteristics for each column of data. Data will be released directly by Dr. Otto's team at Boston University to investigators providing evidence of their institution's approval for planned analyses of the data.
Supporting Information: Study Protocol, SAP
Time Frame: Within one year of completion (publication) of the primary Aims for this project,

REFERENCES:
- [Derived] Otto MW, Zvolensky MJ, Rosenfield D, Hoyt DL, Witkiewitz K, McKee SA, Bickel WK, Smits JAJ. A randomized controlled trial protocol for engaging distress tolerance and working memory to aid smoking cessation in low socioeconomic status (SES) adults. Health Psychol. 2020 Sep;39(9):815-825. doi: 10.1037/hea0000858. PMID 32833483

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were three reasons why enrolled participants were not randomized to study groups: lost contact (3 participants), subject withdrew themselves (2 participants) and issues with commuting to study site (1 participant). Six participants dropped out prior to randomization.
Period: Overall Study
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Started (Participants that were enrolled and randomized to study groups.) | 8 | 8 | 8
V1 (Intervention visit 1 completed.) | 8 | 7 | 7
V2 (Intervention visit 2 completed) | 8 | 7 | 5
V3 (Intervention visit 3 completed) | 6 | 6 | 5
V4 (Intervention visit 4 completed) | 6 | 6 | 5
V5 (Intervention visit 5 completed) | 6 | 6 | 5
V6 (Intervention visit 6 completed) | 6 | 6 | 5
SSA (1-week Post-Intervention Smoking Context- Standard smoking assessment (SSA) completed) | 6 | 6 | 5
DWA (1week+2days Post-Intervention Deprivation Context- Deprivation window assessment (DWA) completed) | 6 | 5 (One participant from MT group refused the McKee protocol and dropped out of the study during the DWA visit. Data was collected for some outcome variables during this visit, but not all. This participant's data was not included in the calculation of primary outcome measures.) | 4
PFU (6 week Post-Intervention- Phone follow-up (PFU) completed) | 6 | 5 | 4
Completed | 6 | 5 | 4
Not Completed | 2 | 3 | 4
Not completed — COVID-19 halt to human subjects research | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — Information on participant's date of birth was collected. This date was then compared to the date the study visit took place to calculate the participant's age. Population: Age was calculated from date of birth. One participant in the Mindfulness + IE listed the date of their study visit as DOB, and therefore, we were unable to calculate age.
  years
    number analyzed (Participants) | 8 | 8 | 7 | 23
    (all) | 49.56 (8.31) | 45.63 (13.59) | 47.14 (10.92) | 47.46 (10.77)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Reported Gender: Male | 6 | 7 | 4 | 17
  Reported Gender: Female | 2 | 1 | 3 | 6
  Reported Gender: Transgender | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 5
  Not Hispanic or Latino | 6 | 7 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 4 | 13
  White | 3 | 2 | 1 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 8 | 24
Fagerstrom Test for Nicotine Dependence (FTND) [Mean (Standard Deviation); unit: units on a scale] — Self-report assessment designed to assess gradations in cigarette dependence. All 6 items are summed to compute a composite total score. Scores range from 0 to 10. Scores of 1-2 indicate low dependence on nicotine. Scores of 3-4 indicate a low to moderate dependence on nicotine. Scores of 5-7 indicate a moderate dependence on nicotine. Scores of 8+ indicate a high dependence on nicotine.
  units on a scale | 3.13 (1.73) | 4.37 (2.77) | 5.13 (1.13) | 4.21 (2.08)
Smoking Urges (QSU) [Mean (Standard Deviation); unit: units on a scale] — Self-report assessment used to characterize smoking behavior. 10 items are rated on a scale from 1 (strongly disagree) to 7 (strongly agree). Items are summed to create a composite total score. Scores range from 10 to 70. Higher scores indicated stronger smoking urges.
  units on a scale | 36.75 (14.97) | 36.75 (14.72) | 38.75 (13.38) | 37.42 (15.79)
Executive Function (BRIEF A) [Mean (Standard Deviation); unit: units on a scale] — Baseline levels of behavioral regulation was assessed with the global executive composite raw score from the Behavioral Rating Inventory of Executive Function-Adult (BRIEF-A). The measure utilizes a standardized self-report form and standardized scoring instructions. Items are summed to create the Global Executive Composite (GEC) raw score, reported here. Scores on the GEC range from a minimum of 70 to a maximum of 210. Higher scores indicate more negative self-evaluation of one's executive functioning.
  units on a scale | 91.63 (16.19) | 101.12 (27.72) | 111.75 (26.03) | 101.50 (24.29)
Psychological Distress (Kessler K6+) [Mean (Standard Deviation); unit: units on a scale] — Baseline levels of psychological distress were assessed with the Kessler Psychological Distress Scale (K6+). All 6 items are summed to compute a composite total score. Scores range from 0 to 24. Higher scores indicate more severe mental illness/distress, with scores of 13-24 indicating a serious clinical mental illness.
  units on a scale | 2.00 (2.00) | 5.13 (4.55) | 9.00 (6.70) | 5.38 (5.45)

OUTCOME MEASURES:

1. Primary Outcome: Negative Affect
Description: PANAS-State Negative was used to assess the mechanistic outcome of Negative Affectivity/Stress. Items from the negative subscale are summed to create a total score. Scores can range from 10-50, with lower scores representing lower levels of negative affect.
Time Frame: 1-week Post-Intervention Smoking Context
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 6 | 5
score on a scale | 11.33 (1.21) | 12.67 (3.56) | 24.20 (9.18)

2. Primary Outcome: Negative Affect/Withdrawal
Description: Wisconsin Smoking Withdrawal Scale (WSWS) was used to assess withdrawal symptoms. Some items are reversed scored and the average of all items is calculated. Scores range between 0 and 4, with higher scores indicating stronger withdrawal symptoms.
Time Frame: 1-week Post-Intervention Smoking Context
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 6 | 5
score on a scale | 1.81 (0.61) | 1.84 (0.19) | 2.24 (0.46)

3. Primary Outcome: N-Back Task
Description: Adaptive N-Back task is a continuous performance task that was administered on the computer. It was used to assess working memory capacity. The participant is present with a series of stimuli and asked to identify when the current stimulus matches the one from n back steps prior. For the current task, n was equal to 2. As such, the score reported is the total number of correct trials form the 2-back condition of the computer task. Higher scores indicate better working memory capacity. Participant completed 20 trials. The task was administered online and can be found at: https://measures.scienceofbehaviorchange.org/measuredetails/d4a117c9-e5d8-41a0-8227-ac570a60f89f.
Time Frame: 1-week Post-Intervention Smoking Context
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 6 | 5
score | 113.00 (84.43) | 63.17 (53.11) | 69.00 (101.16)

4. Primary Outcome: Spatial Span
Description: The mechanistic outcome of working memory was assessed by summing the number of correct trials on the backwards spatial span task. The spatial span task was administered via computer. On each trial, participants see an array of geometric shapes (white squares) on the screen. The squares change from white to a different color in a sequence with variable orders and colors. At the end of the list sequences, the participants attempt to recall the squares in the reverse order that they changed color. The difficulty on each trial is increased by varying the number of boxes from two (easiest) to nine (hardest). The maximum number of boxes correctly recalled is the outcome measure. Higher numbers of boxes recalled indicates increased working memory capacity. The task was administered online from the SOBC Repository and is available at: https://scienceofbehaviorchange.org/measures/spatial-span-task/.
Time Frame: 1-week Post-Intervention Smoking Context
Measure: Mean (Standard Deviation); unit: number of correct trials
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 6 | 5
number of correct trials | 5.17 (0.98) | 5.33 (0.52) | 5.20 (0.84)

5. Primary Outcome: Digit Span
Description: The mechanistic outcome of working memory was assessed by taking the longest span of correct answers on the backwards digit span task. The digit span task was administered via computer. On each trial, participants are presented with lists of digits 1 at a time on the screen. At the end of each list, participants attempt to recall the digits in reverse ordered they appeared by typing them in. After each successfully completed trial, the number of digits in the list is increased by 1 for the next trial. After a failed trial, the number of digits remains the same for the next trial. The task ends when the participant makes errors for two trails in a row for a given digit span. The maximum number of digits correctly recalled is the outcome measure. Higher numbers (more digits) indicated increased working memory capacity. The task was administered online from the SOBC Repository and is available at: https://scienceofbehaviorchange.org/measures/digit-span-task/.
Time Frame: 1-week Post-Intervention Smoking Context
Measure: Mean (Standard Deviation); unit: longest span of correct answers
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 6 | 5
longest span of correct answers | 5.83 (0.41) | 5.33 (2.06) | 4.20 (1.30)

6. Primary Outcome: Anxiety Sensitivity
Description: The mechanistic outcome of distress tolerance was assessed with the Anxiety Sensitivity Index (ASI 3). Items on this scale are summed, with scores ranging from 0-72. Higher scores indicate worse outcome.
Time Frame: 1-week Post-Intervention Smoking Context
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 6 | 5
score on a scale | 8.00 (12.96) | 13.67 (10.41) | 22.20 (9.18)

7. Primary Outcome: Mirror-Tracing Persistence Task
Description: The mechanistic outcome of behavioral distress tolerance was assessed with the mirror-tracing persistence task. The task measures how long the participant persists in completing the tracing tasks. Longer times are indicative of better behavioral stress tolerance capacity.
Time Frame: 1-week Post-Intervention Smoking Context
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 6 | 5
seconds | 93.31 (68.86) | 255.85 (291.89) | 136.11 (112.22)

8. Primary Outcome: Negative Affect
Description: as for outcome 1
Time Frame: 1week+2days Post-Intervention Deprivation Context
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 5 | 4
score on a scale | 10.33 (0.82) | 14.40 (6.12) | 21.25 (6.40)

9. Primary Outcome: Negative Affect/Withdrawal
Description: as for outcome 2
Time Frame: 1week+2days Post-Intervention Deprivation Context
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 5 | 4
score on a scale | 1.73 (0.67) | 1.89 (0.17) | 2.06 (0.27)

10. Primary Outcome: N-Back Task
Description: as for outcome 3
Time Frame: 1week+2days Post-Intervention Deprivation Contex
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 5 | 4
score | 103.33 (99.49) | 75.20 (52.79) | 11.50 (8.96)

11. Primary Outcome: Spatial Span
Description: as for outcome 4
Time Frame: 1week+2days Post-Intervention Deprivation Contex
Measure: Mean (Standard Deviation); unit: number of correct trials
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 5 | 4
number of correct trials | 5.17 (0.98) | 5.60 (0.55) | 4.50 (0.58)

12. Primary Outcome: Digit Span
Description: as for outcome 5
Time Frame: 1week+2days Post-Intervention Deprivation Context
Measure: Mean (Standard Deviation); unit: longest span of correct answers
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 5 | 4
longest span of correct answers | 6.33 (1.03) | 5.60 (1.82) | 4.25 (0.96)

13. Primary Outcome: Anxiety Sensitivity
Description: as for outcome 6
Time Frame: 1week+2days Post-Intervention Deprivation Contex
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 5 | 4
score on a scale | 6.67 (10.63) | 14.40 (11.76) | 17.50 (19.05)

14. Primary Outcome: Mirror-Tracing Persistence Task
Description: as for outcome 7
Time Frame: 1week+2days Post-Intervention Deprivation Context
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 5 | 4
seconds | 65.67 (39.35) | 137.83 (64.43) | 47.91 (55.49)

15. Secondary Outcome: McKee Protocol Delay Until Smoking
Description: Degree of delay (in minutes) until smoking in the McKee protocol. The number of minutes the participant went during the delay period without smoking is reported. If the participant did not smoke at all during the delay period, the value is 50.
Time Frame: 1week+2days Post-Intervention Deprivation Context
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 6 | 6 | 4
minutes | 45.83 (10.21) | 46.17 (9.39) | 27.00 (26.76)

16. Secondary Outcome: McKee Protocol Number of Cigarettes Smoked
Description: Number of cigarettes smoked in the 60 minute self-administration session. No value is entered if the participant did not smoke a cigarette during the session at all. Otherwise, the number reported is the number of cigarettes the participant smoked during the session.
Time Frame: 1week+2days Post-Intervention Deprivation Context
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 3 | 3 | 1
cigarettes | 1.00 (0.00) | 2.00 (1.73) | 2.00 (NA) — Data was only collected on one participant, therefore a standard deviation cannot be calculated.

17. Secondary Outcome: Smoking Topography-1
Description: Puff CO volume. During administration of this assessment, there was equipment failure. For this reason, no participants had valid data collected or analyzed for this measure.
Time Frame: 1week+2days Post-Intervention Deprivation Context
Population: During administration of this assessment, there was equipment failure. For this reason, no participants had valid data collected or analyzed for this measure.
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Smoking Topography-2
Description: as for outcome 17
Time Frame: 1week+2days Post-Intervention Deprivation Context
Population: During administration of this assessment, there was equipment failure. No participants had valid data collected or analyzed for this measure.
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Smoking Topography-3
Description: Inter-puff interval. During administration of this assessment, there was equipment failure. For this reason, no participants had valid data collected or analyzed for this measure.
Time Frame: 1week+2days Post-Intervention Deprivation Context
Population: as for outcome 18
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time the participant was enrolled at week 0 until the completion of the follow up phone call at week 11.
Arm/Group | Wellness Education Control Condition | Mindfulness Training (MT) | Mindfulness Training Plus IE (MT+IE)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Early termination of the study due to the COVID-19 shut down of human subjects research led to a small number of participants enrolled in the study and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT03565497/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT03565497/SAP_001.pdf